CLINICAL TRIAL: NCT05287347
Title: Prospective Multicenter Observational Study for Validation of a Pancreatic Cancer Risk Model and Assessment of the Predictive Value of Blood Biomarkers in a High-risk Cohort
Brief Title: Panc CA Risk Model & Biomarker Testing In High-Risk Cohort
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Limor Appelbaum, Principal Investigator, Beth Israel Deaconess Medical Center
Other Study IDs: 21-490
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic Adenocarcinoma
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Specimen collection:
  1. Tumor markers CEA, CA 19-9: 2 ml blood for will be collected in a serum separator tube, processed at each institution and serum stored locally in -80C freezers. Samples will be shipped in batches every 2 months to BIDMC for tumor marker analysis, and results recorded and blinded until the end of the study collection period.
  2. Serum glycomics: 0.5 cc of blood will be collected in sterile Vacutainer tubes. Serum will be separated and aliquoted in 50 microliters aliquots, and frozen at -80C, for up to 3 years.
  3. ctDNA, 20 cc of blood will be collected from patients in specialized tubes to stabilize the leukocytes and avoid contamination by genomic DNA. Samples will be processed within 48 hours to separate plasma, which will be frozen for batch analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prospective: Blood specimens will be obtained for the model-assigned high risk cohort at each collaborating HCO, over two years of recruitment period. Data of each participant will be electronically followed for observation of outcome measures for up to 3 years.
  Interventions: Diagnostic Test: Blood Specimen

INTERVENTIONS:
Diagnostic Test: Blood Specimen — Blood samples will be collected from study participants at one time-point in the study, for the following:
  1. tumor markers CEA and CA 19-9: 2 ml blood will be collected.
  2. glycomics: 0.5 cc blood will be collected
  3. ctDNA: 20 cc blood will be collected

SUMMARY:
The purpose of this study is to test a double screening strategy for pancreatic cancer, based on a model developed using patient medical records. Investigators would also like to test whether adding specific blood tests, can further help identify people who have a higher risk of pancreatic cancer than the general population, and would benefit from imaging in order to detect cancer early.

DETAILED DESCRIPTION:
This research aims to identify people who have a higher risk of pancreatic cancer than the general population, by testing a double-screening strategy for pancreatic cancer. The purpose is to allow early detection of cancer, which potentially leads to cure.

The double-screening will include a computer-based model developed using clinical data from medical records, and three different blood tests for early detection of pancreatic cancer.

Participation in this study involves having medical records followed up for up to three years, and a single donation of blood specimens.

- This is a Combined Retrospective and Prospective Review:

* The first part of the study, involves collection of retrospective data from Electronic Health Record database (for the 3 collaborating HCOs) in order to deploy our EHR model, so that a high-risk group for pancreatic cancer can be identified. All individuals stratified into low, intermediate or high risk groups by the model, will be prospectively, electronically followed to assess outcome.
* The second stage is prospective, and involves requesting biological specimen donations from participants identified as high-risk, for biomarker testing. The prospective "observation period" is up to 3 years (depending on each subject's index date at retrospective recruitment and outcome). Biological specimens will be collected during the prospective "observation period,"

ELIGIBILITY:
Inclusion Criteria:

* Study population for part 1 of study:

  -- Inclusion criteria: i) Male and females age >= 50 years; ii) at least one clinical visit to an outpatient clinic of the HCO, within the last year, before the study start date.
* Study population for part 2 of study:

  * i) model-assigned high-risk subjects; ii) Male and females age >= 50 years; iii) at least one clinical visit to an outpatient clinic of the HCO, within the last year, before the study start date

Exclusion Criteria:

* Exclusion Criteria for part 1 of study:

  * Personal history of PDAC or current PDAC
  * Age below 50.
* Exclusion Criteria for part 2 of study

  * model-assigned low or intermediate risk subjects
  * Personal history of PDAC or current PDAC
  * Age below 50.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population for part 1 of study:
  * Inclusion criteria: i) Male and females age >= 50 years; ii) at least one clinical visit to an outpatient clinic of the HCO, within the last year, before the study start date.
    - Study population for part 2 of study:
  * i) model-assigned high-risk subjects
  * ii) Male and females age >= 50 years;
  * iii) at least one clinical visit to an outpatient clinic of the HCO, within the last year, before the study start date
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Incident PDAC during the 3-year study observation period | 3 Years
  The diagnosis of PDAC will be determined by ICD code (ICD10 codes C25.X, excluding C25.4), tumor registry records or pathology reports

SECONDARY OUTCOMES:
Timing of incident PDAC occurrence | 3 Years
  time from index date to diagnosis
Tumor stage at PDAC diagnosis | 3 Years
  stage at diagnosis per tumor registry/pathology report

CONTACTS AND LOCATIONS:
Overall Officials: Limor Appelbaum, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu